CLINICAL TRIAL: NCT00741078
Title: Additive Beneficial Effects of Atorvastatin Combined With Amlodipine In Treatment of Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Model: Crossover | Purpose: Treatment
Other Study IDs: GMC-200504
Record Dates: First submitted 2008-08-20; First posted 2008-08-26 (Estimated); Last update posted 2008-08-29 (Estimated); Status verified 2008-08

CONDITIONS: Hypertension
Keywords: endothelial; function; insulin; sensitivity
MeSH Terms: conditions — Hypertension; Insulin Resistance; Hypersensitivity | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- atorvastatin, amlodipine (Experimental)
  Interventions: Drug: statin, amlodipine

INTERVENTIONS:
Drug: statin, amlodipine

SUMMARY:
The investigators hypothesized combination therapy would be superior to monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension

Exclusion Criteria:

* Chronic renal disease
* Severe hypertension

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-12; Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Gil Medical Center, Incheon, South Korea